CLINICAL TRIAL: NCT04931589
Title: A Multicentre Study of Intraoperative Body Temperature Changes in Patients Undergoing Thoracoscopic Radical Surgery for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-004
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-01

CONDITIONS: Body Temperature Protection; Video-assisted Thoracic Surgery; Lung Cancer; Nursing Caries
Keywords: Thoracoscopy; Lung cancer; Surgery; Body temperature; Nursing; multicenter
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the "Curve of Intraoperative Body Temperature Change in Patients with VATS Surgery" was taken as the main research content to retrospectively analyze the intraoperative body temperature and its change rules of patients who met the research conditions, and draw a trend curve, namely, the curve of body temperature change.Taking "time" as the independent variable and "body temperature" as the dependent variable, the correlation between the two was statistically analyzed.Through the development of the body temperature change curve, we can further understand the phenomenon that the body temperature of patients undergoing VATS surgery changes with the progress of surgery, and longitudinal understand the change trend and the general rule of the body temperature change.The results can provide a basis for clinical development of scientific preoperative evaluation plan, hypothermia prevention strategy and intraoperative intervention plan.

DETAILED DESCRIPTION:
Lung cancer is a common malignant tumor. With the increasingly serious air pollution and the arrival of the aging society, the prevalence of lung cancer is increasing year by year.According to the Globocan 2018 Cancer Report, published 2018 by the International Agency for Research on Cancer (IARC) of the World Health Organization,Lung cancer accounted for 11.6% of new cases and 18.4% of deaths from malignancies globally in 2018, ranking first among malignancies.As the mainstream surgical treatment of lung cancer, video-assisted thoracic surgery (VATS) has many advantages such as less trauma and rapid recovery of patients, and has become one of the preferred methods for the treatment of lung cancer, especially early lung cancer.It has been widely used at home and abroad.However, with the more and more extensive development of VATS surgery, the phenomenon of intraoperative hypothermia in patients is relatively common clinically.The study results of Cywinski et al. showed that the rate of hypothermia after thoracoscopic surgery could reach 50%.Intraoperative hypothermia can lead to adverse effects such as increased cardiovascular events, coagulation dysfunction, prolonged wound recovery time, increased risk of wound infection, immune system suppression, and slow drug metabolism [7].

Perioperative hypothermia means that the body's core body temperature is less than 36℃ due to various reasons during the perioperative period, also known as perioperative unexpected hypothermia or unplanned perioperative hypothermia.Perioperative hypothermia can be caused by any factor that may affect thermoregulation.Risk factors affecting thermoregulation mainly include patient anesthesia factors, self factors, surgical factors, environmental factors, etc. [13].Operation when the room temperature is too low, inadequate coverage and other factors leading to excessive heat loss surgery (room temperature as a given intravenous fluids and rinses, evaporation of the skin disinfectant, etc.), lead to the low temperature of unplanned, patients not only affect the function of blood coagulation, lead to increased perioperative blood loss, also can increase the risk of cardiovascular events, and can suppress the immune function,It can lead to postoperative infection and even more serious adverse outcomes.Intraoperative hypothermia involved in this study includes perioperative hypothermia, which is an important clinical manifestation of perioperative hypothermia.It is found in clinical practice that the proportion of intraoperative hypothermia in patients undergoing VATS surgery is high, which is closely related to the specific surgical position and surgical site.

Current studies on intraoperative hypothermia in patients undergoing VATS surgery [15-16] mainly focus on the comparison of intervention methods, including the selection of intervention methods, the effect comparison of heating equipment, or the effect comparison of heating sites.However, there has been no in-depth study on the specific changes of body temperature and the trend of body temperature changes during VATS surgery.At the same time, the intervention time point for intraoperative hypothermia is mainly judged by clinical experience, and there is a lack of support from objective data studies.Clinical observation shows that the changes of body temperature in patients undergoing VATS surgery are not a straight line, nor a simple arc, but a curve that changes continuously with the operation time.

In this study, the "Curve of Intraoperative Body Temperature Change in Patients with VATS Surgery" was taken as the main research content to retrospectively analyze the intraoperative body temperature and its change rules of patients who met the research conditions, and draw a trend curve, namely, the curve of body temperature change.Taking "time" as the independent variable and "body temperature" as the dependent variable, the correlation between the two was statistically analyzed.Through the development of the body temperature change curve, we can further understand the phenomenon that the body temperature of patients undergoing VATS surgery changes with the progress of surgery, and longitudinal understand the change trend and the general rule of the body temperature change.The results can provide a basis for clinical development of scientific preoperative evaluation plan, hypothermia prevention strategy and intraoperative intervention plan.Moreover, it can further study the influence of various factors, such as surgical factors, anesthesia factors and patients' own factors, on the temperature change curve, so as to provide a basis for clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* ① Endoscopic radical resection of lung cancer was performed with a single or porous approach.② Continuous monitoring of nasopharyngeal temperature was recorded during the whole operation (the system automatically recorded once every 5min);③ The preoperative basal metabolism was normal, and the basal body temperature was 36.5℃<T0<37.5℃ (the preoperative average body temperature in hospital);(4) total subvenous tracheal intubation anesthesia;

Exclusion Criteria:

* Patients with the minimum intraoperative temperature monitoring data >36.0℃;Cases with warm intervention immediately after the start of surgery;Patients undergoing combined surgery for other types or organs;Intraoperative monitoring of body temperature was discontinuous or abnormal (monitoring catheter was accidentally pulled out, etc.);Intraoperative endoscopic change cases;Other cases that do not meet the requirements of the study, such as individual data anomalies or cases that are far more specific than the general cases (the cases themselves are special or caused by human recording errors).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All surgical patients from Vast
Sampling Method: Non-Probability Sample
Enrollment: 2156 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Body temperature | Estimated time for each operation is 60-240 minutes
  Temperature per 5 minutes during the operation

CONTACTS AND LOCATIONS:
Overall Officials: lina Yu, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No